CLINICAL TRIAL: NCT01352299
Title: Comparison of Visualisation of Laryngeal Inlet and Ease of Intubation With Different Laryngoscope Blades.
Brief Title: Glottic Visualization & Ease of Intubation With Different Laryngoscope Blades
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Dr Atul P Kulkarni, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Akulkarni2
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Tracheal Intubation Morbidity
Keywords: Macintosh laryngoscope blade; MacCoy laryngoscope blade; Miller laryngoscope blade; TrueView laryngoscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Macintosh (Active Comparator): Laryngoscopy performed with Macintosh Laryngoscope
  Interventions: Device: Macintosh Laryngoscope blade
- McCoy (Active Comparator): Laryngoscopy performed with MacCoy Laryngoscope
  Interventions: Device: MacCoy
- Miller (Active Comparator): Laryngoscopy performed with Miller Laryngoscope
  Interventions: Device: Miller
- TrueView (Active Comparator): Laryngoscopy performed with TrueView Laryngoscope
  Interventions: Device: TrueView

INTERVENTIONS:
Device: Macintosh Laryngoscope blade — Laryngoscopy performed with Macintosh Laryngoscope
  Other Names: Conventional Curved laryngoscope blade
  Arms: Macintosh
Device: MacCoy — Laryngoscopy performed with MacCoy Laryngoscope
  Other Names: Curved laryngoscope blade with a hinged tip
  Arms: McCoy
Device: Miller — Laryngoscopy performed with Miller Laryngoscope
  Other Names: Conventional Straight laryngoscope blade
  Arms: Miller
Device: TrueView — Laryngoscopy performed with TrueView laryngoscope
  Other Names: Straight blade with prism
  Arms: TrueView

SUMMARY:
Orotracheal intubation the commonest method used to secure and maintain airway during anaesthesia. A variety of methods are available for orotracheal intubation such as digital or tactile method, use of lighted orotracheal intubating stylet, use of intubating LMA (which is becoming increasing popular, particularly in cased of anticipated difficult intubation), fibreoptic endoscopic orotracheal intubation (also used when a difficulty is predicted), and conventional and most common method, direct laryngoscopy. Orotracheal intubation is most commonly achieved after visualization of laryngeal inlet with direct laryngoscopy following induction of general anaesthesia and muscle relaxation achieved by administration of a muscle relaxant.

Due to the hazards seen with failed intubation, anaesthetists are also on the lookout for techniques which will improve visualization of the laryngeal inlet, i.e. glottis. View obtained during laryngoscopy can be classified in a variety of ways such as Cormack Lehane grading, the percentage of glottic opening (POGO Score)Literature suggests that straight blade gives better glottic visualization while tracheal intubation is easier with the curved blade. We therefore wanted to compare the Macintosh and Miller laryngoscope blades in terms of visualization of Laryngeal inlet and ease of intubation in patients with normal predicted intubation. We also compared the McCoy blade, a modified curved blade, and the Trueview Laryngoscope, which incorporates a prism in a straight blade, for glottic view and ease of intubation.

DETAILED DESCRIPTION:
This prospective observational study was conducted after obtaining approval from the Institutional Review board of our institute. One hundred and twenty adult patients were included who had given written informed consent. These patients were ASA I or II, between 18-70 yrs of age, were undergoing elective oncosurgery procedure under general anaesthesia requiring endotracheal intubation. Patinets were excluded if they refused consent, were pregnant, had potential difficult mask ventilation and /or anticipated difficult intubation or had pathology in neck, upper respiratory tract and upper alimentary tract. A detailed routine pre-anaesthetic check-up was performed and routine laboratory investigations were done. The patients were randomly divided in four groups of 30 each per laryngoscope blade. Group 1: Macintosh Group Group 2: McCoy's Group Group 3 Miller Group and Group 4: TrueView Group. : included 30 patients.

In the operating room, patients' medical history was again confirmed in brief before subjecting the patient to anaesthesia. Demographic data such as age, sex and weight of the patient was noted. Pulse oximeter, electrocardiograph, capnography and automated non-invasive blood pressure were used for monitoring. Airway assessment was done clinically using Samsung and Young's modification of the Mallampati classification for oropharyngeal view. The patient was asked to assume sitting position, open the mouth maximally, and protrude the tongue but not to phonate. Visibility of the oral and pharyngeal structures was then classified by an observer sitting at the same level as the patient.

Class I: Soft palate,fauces,uvula,pillars visible Class II: Soft palate,fauces,portion of uvula visible Class III: Soft palate,base of uvula visible Class IV : Only hard palate visible A Doughnut-shaped pillow and hard sponge square pillow, totalling about 7 cm in height, was placed under the head of the patient. The patient was preoxygenated with 100% oxygen for three minutes. Anaesthesia was then induced with 1-3 mg/kg of Propofol or thiopentone sodium 5 mg/kg, fentanyl 2 µg/kg. Feasibility of ventilation with a face mask was checked prior to injection of non-depolarising muscle relaxant. After ventilation was confirmed a vecuronium was administered and the patient was ventilated with isoflurane 0.5-1% in a 50:50 mixture of O2 and N2O for 3 minutes then ventilated for 1 minute with 100% O2. Then laryngoscopy and tracheal intubation accomplished with the selected laryngoscope blade. The laryngoscopy and intubation were carried out by a single anaesthesiologist who had trained with all laryngoscope blades till he had obtained sufficient familiarity all four laryngoscope blades. We studied following aspects during tracheal intubation.

Visualization of laryngeal inlet: This was graded using Cormack Lehane Grades:

Grade 1: complete glottis visible Grade 2: anterior glottis not seen Grade 3: epiglottis seen but not glottis Grade 4: epiglottis not seen

Ease of intubation: This was graded as follows:

Grade 1: Intubation easy Grade 2: Intubation requiring an increased anterior lifting force and assistance to pull the right corner of the mouth upwards to increase space Grade 3: Intubation requiring multiple attempts and a curved stylet Grade 4: Failure to intubate with the assigned laryngoscope Number of attempts: We noted the number of attempts needed for intubation with that particular blade in each patient.

Requirement of external laryngeal manipulation: Classified as Grade 1: No requirement of external laryngeal manipulations and Grade 2: Requirement of external laryngeal manipulation.

Statistical analysis: Demographic data, Mallampatti Classification and other variables were compared using the Chi Square test. A p value of > 0.05 was taken to assume statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the age group of 18-70 yrs
* Patients with ASA grade I and II
* Undergoing surgery under general anaesthesia requiring endotracheal intubation.

Exclusion Criteria:

* Patient's refusal for consent for study.
* Patients less than 18 years and more than 70years of age.
* Pregnant patients
* Patients with difficult mask ventilation and /or anticipated difficult intubation
* Patients with pathology in neck, upper respiratory tract and upper alimentary tract.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Visualization of glottis and Ease of Intubation | During Laryngoscopy and intubation average time 1 minute
  Visualization of laryngeal inlet:
  Grade 1: complete glottis visible Grade 2: anterior glottis not seen Grade 3: epiglottis seen but not glottis Grade 4: epiglottis not seen
  Ease of intubation:
  Grade 1: Intubation easy Grade 2: Intubation requiring an increased anterior lifting force and assistance to pull the right corner of the mouth upwards to increase space Grade 3: Intubation requiring multiple attempts and a curved stylet Grade 4: Failure to intubate with the assigned laryngoscope

CONTACTS AND LOCATIONS:
Overall Officials: Atul P Kulkarni, MD Anaes, Principal Investigator — Professor Tata Memorial Hospital
Locations (1):
- Tata Memorial Hopsital, Mumbai, Maharashtra, India